CLINICAL TRIAL: NCT03505320
Title: A Phase 2 Study of Zolbetuximab (IMAB362) as Monotherapy and in Combination With Chemotherapy and/or Immunotherapy in Subjects With Metastatic or Locally Advanced Unresectable Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma and Locoregional Gastric or GEJ Adenocarcinoma Whose Are Claudin (CLDN) 18.2 Positive
Brief Title: A Study of Zolbetuximab (IMAB362) in Adults With Gastric Cancer
Acronym: ILUSTRO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8951-CL-0103; 2017-002566-50 (EudraCT Number); jRCT2080225325 (Registry Identifier: jRCT); 2024-511649-21-00 (Registry Identifier: CTIS (EU))
Expanded Access: NCT06048081 (Available)
Record Dates: First submitted 2018-03-29; First posted 2018-04-23 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Pharmacokinetics of Zolbetuximab; Gastric Cancer; Gastro-esophageal Junction (GEJ) Cancer; Pharmacokinetics of Oxaliplatin; Pharmacokinetics of Fluorouracil Bolus (5-FU)
Keywords: zolbetuximab; oxaliplatin; fluorouracil; docetaxel; claudiximab; IMAB362; Gastro-Esophageal Junction cancer; locoregional gastric cancer; Pembrolizumab; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms | interventions — zolbetuximab; Oxaliplatin; Leucovorin; Fluorouracil; pembrolizumab; Nivolumab; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants will be enrolled to receive zolbetuximab as monotherapy or in combination with mFOLFOX6 (with or without Nivolumab) and in combination with pembrolizumab and in combination with FLOT in an unblinded fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- zolbetuximab (Cohort 1A) (Experimental): Participants will be treated with zolbetuximab on a 21-day cycle in which zolbetuximab will be administered as a single agent every 3 weeks until disease progression, toxicity requiring cessation, start of another anti-cancer treatment or other treatment discontinuation criteria are met.
  Interventions: Drug: zolbetuximab
- mFOLFOX6 plus zolbetuximab (Cohort 2) (Experimental): Participants will be treated with zolbetuximab and mFOLFOX6 on a 42-day cycle in which zolbetuximab is administered on days 1 and 22, and mFOLFOX6 is administered on days 1, 15 and 29; however, for the first cycle, zolbetuximab will be administered on day 3 (instead of day 1) to allow for pharmacokinetic collection. Participants will receive up to 12 mFOLFOX6 treatments (4 cycles). Beginning at cycle 5, participants may continue on 5-FU and leucovorin or folinic acid along with zolbetuximab for the remainder of the study per investigator's discretion. mFOLFOX6 treatment includes oxaliplatin: intravenous [IV] infusion, leucovorin: IV infusion, fluorouracil bolus: IV bolus, fluorouracil infusion: continuous IV infusion.
  Interventions: Drug: zolbetuximab; Drug: oxaliplatin; Drug: leucovorin; Drug: fluorouracil; Drug: folinic acid
- Pembrolizumab plus zolbetuximab (Cohort 3A) (Experimental): Participants will be treated with zolbetuximab and pembrolizumab on a 21-day cycle. Loading dose of zolbetuximab will be administered at cycle 1, day 1 followed by maintenance dose of zolbetuximab once every 3 weeks (Q3W). Pembrolizumab will be administered to 3 to 6 subjects at a intravenously on day 1 of every 21-day cycle and will be infused 1 hour after the zolbetuximab infusion is completed. Tolerability and safety of zolbetuximab in combination with pembrolizumab will be evaluated during the 3-week dose-limiting toxicity (DLT) assessment period. If this cycle 1 dose is not tolerable, a lower dose of zolbetuximab in combination with pembrolizumab will subsequently be evaluated.
  Interventions: Drug: zolbetuximab; Drug: Pembrolizumab
- Zolbetuximab in combination with mFOLFOX6 and nivolumab (Cohort 4A/4B) (Experimental): Participants will be treated with zolbetuximab and mFOLFOX6, nivolumab on a 42-day cycle. Cohort 4A: Loading dose of zolbetuximab in combination with nivolumab and mFOLFOX6 on cycle 1 day 1, followed by zolbetuximab in combination with nivolumab and mFOLFOX6 q2w [days 15 and 29] (1 cycle = 6 weeks). Tolerability and safety of zolbetuximab in combination with nivolumab, mFOLFOX6 will be evaluated during the 3-week DLT assessment period. If cycle 1 dose is not tolerable, a lower dose of dose zolbetuximab in combination with nivolumab and mFOLFOX6 will be subsequently evaluated. Cohort 4B: Subjects will be treated with the combination of zolbetuximab, mFOLFOX6 and nivolumab at the dose deemed tolerable in Cohort 4A. Subjects will receive up to 12 mFOLFOX6 treatments (4 cycles). For Cohorts 4A and 4B, beginning at cycle 5, subjects may continue on 5-FU and leucovorin or folinic acid along with zolbetuximab and nivolumab for the remainder of the study per investigator's discretion.
  Interventions: Drug: zolbetuximab; Drug: oxaliplatin; Drug: leucovorin; Drug: fluorouracil; Drug: folinic acid; Drug: nivolumab
- Zolbetuximab in combination with FLOT (Cohort 5) (Experimental): Participants will be treated with zolbetuximab & FLOT for a total of eight 2-week cycles. 4 cycles preoperatively & 4 cycles postoperatively 6-12 weeks after surgery.
  Preoperative: Participants will receive zolbetuximab loading dose on cycle 1 day 1, followed by FLOT on cycle 1 day 2. For cycles 2-4, participants may receive zolbetuximab maintenance dose in combination with FLOT, dosed on day 1 of each cycle. However, dosing may be split over 2 days with zolbetuximab administration on day 1 & FLOT on day 2.
  Post operative: Participants will receive zolbetuximab loading dose on cycle 5 day 1, followed by FLOT on cycle 5 day 2. For cycles 6-8, participants may receive zolbetuximab maintenance dose in combination with FLOT, dosed on day 1 of each cycle. However, dosing may be split over 2 days with zolbetuximab administration on day 1 and FLOT on day 2. For participants who experience a DLT during preoperative treatment on the loading dose, the postoperative loading dose may be lowered.
  Interventions: Drug: zolbetuximab; Drug: oxaliplatin; Drug: leucovorin; Drug: fluorouracil; Drug: folinic acid; Drug: Docetaxel

INTERVENTIONS:
Drug: zolbetuximab — Zolbetuximab will be administered as a minimum 2-hour IV infusion.
  Other Names: IMAB362
Drug: oxaliplatin — Oxaliplatin will be administered as a 2-hour IV infusion.
  Arms: Zolbetuximab in combination with FLOT (Cohort 5); Zolbetuximab in combination with mFOLFOX6 and nivolumab (Cohort 4A/4B); mFOLFOX6 plus zolbetuximab (Cohort 2)
Drug: leucovorin — Leucovorin will be administered as a 2-hour IV infusion.
  Arms: Zolbetuximab in combination with FLOT (Cohort 5); Zolbetuximab in combination with mFOLFOX6 and nivolumab (Cohort 4A/4B); mFOLFOX6 plus zolbetuximab (Cohort 2)
Drug: fluorouracil — Fluorouracil will be administered as IV bolus over 5 to 15 minutes and continuous IV infusion over 46 to 48 hours or per institutional guidelines.
  Arms: Zolbetuximab in combination with FLOT (Cohort 5); Zolbetuximab in combination with mFOLFOX6 and nivolumab (Cohort 4A/4B); mFOLFOX6 plus zolbetuximab (Cohort 2)
Drug: Pembrolizumab — Pembrolizumab will be administered intravenously over 30 minutes.
  Arms: Pembrolizumab plus zolbetuximab (Cohort 3A)
Drug: folinic acid — Folnic acid will be administered as a 2-hour IV infusion.
  Arms: Zolbetuximab in combination with FLOT (Cohort 5); Zolbetuximab in combination with mFOLFOX6 and nivolumab (Cohort 4A/4B); mFOLFOX6 plus zolbetuximab (Cohort 2)
Drug: nivolumab — Nivolumab will be administered intravenously according to institutional standards.
  Arms: Zolbetuximab in combination with mFOLFOX6 and nivolumab (Cohort 4A/4B)
Drug: Docetaxel — Docetaxel will be administered as a 1-hour IV infusion.
  Arms: Zolbetuximab in combination with FLOT (Cohort 5)

SUMMARY:
Zolbetuximab is being studied as a treatment for people with cancer in and around the stomach or cancer where the food pipe (esophagus) joins the stomach (gastroesophageal junction cancer). Most people with this type of cancer have a protein called Claudin 18.2 in their tumor. Zolbetuximab is thought to work by attaching to Claudin 18.2 in their tumor. This switches on the body's immune system to attack the tumor.

There is an unmet medical need to treat people with advanced cancer in and around the stomach or gastroesophageal junction cancer. This study will provide more information on zolbetuximab given by itself and in combination with other treatments in adults with advanced stomach or gastroesophageal junction cancer. The study is currently ongoing globally. People in this study will either be treated with zolbetuximab by itself, with zolbetuximab and chemotherapy, with zolbetuximab and a medicine called pembrolizumab, or zolbetuximab with chemotherapy and a medicine called nivolumab.

This study is ongoing, but enrollment in any of the treatment options has been completed. In addition, at this stage of the study, treatment in some of these treatment options has completed.

The main aim of this study is to check how well zolbetuximab controls tumors when given by itself.

Adults with cancer in and around the stomach or gastroesophageal junction cancer can take part. Their cancer is locally advanced unresectable or metastatic and has the CLDN18.2 marker in a tumor sample. Locally advanced means the cancer has spread to nearby tissue. Unresectable means the cancer cannot be removed by surgery.

Metastatic means the cancer has spread to other parts of the body. They may have been previously treated with standard therapies. People cannot take part if they need to take medicines to suppress their immune system, have blockages or bleeding in their gut, have specific uncontrollable cancers such as symptomatic or untreated cancers in the nervous system, have a specific heart condition or infections.

There are different treatments in the study. People who take part will receive just 1 of the treatments.

Treatment will be given in cycles. The treatment is given through a vein; this is called an infusion. Some people with advanced disease will have 1 infusion in 3 week (21-day) cycles. Some people will have several infusions in 6 week (42-day) cycles. Some people with cancer in and around the stomach or gastroesophageal junction who have surgery for their cancer will have a few infusions in 2-week (14-day) cycles. This will happen before and after they have surgery for their cancer.

People may receive chemotherapy for up to 6 months. Some people enrolled to received zolbetuximab and pembrolizumab, may have received pembrolizumab for up to 2 years.

People will visit the clinic on certain days during their treatment; there may be extra visits during the first cycle of treatment. The study doctors will check if people had any medical problems from zolbetuximab and the other study treatments. Also, people in the study will have a health check including blood tests. On some visits they will also have scans to check for any changes in their cancer. Tumor samples will be taken at certain visits with the option of giving a tumor sample after treatment has finished.

People will visit the clinic after they stop treatment. They will be asked about any medical problems and will have a health check including blood tests. After the clinic visits end some people will have a telephone health check every 3 months. The number of visits and checks done at each visit will depend on the health of each person and whether they completed their treatment or not.

DETAILED DESCRIPTION:
This is a study to assess the antitumor activity of zolbetuximab, an Immunoglobulin (IgG1) chimeric monoclonal antibody directed against CLDN18.2, in subjects with recurrent locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma and locoregional gastric or GEJ adenocarcinoma whose tumors are CLDN18.2 positive. For each cohort, the study consists of the following periods: pre-screening; screening; treatment; and follow-up for disease progression (or post-treatment follow-up for disease recurrence, which will be conducted for Cohort 5). In addition, there will be a survival follow-up period for Cohorts 1A, 4B, and 5 participants only. Tolerability of zolbetuximab in combination with pembrolizumab in Japanese participant(s) will be evaluated in Cohort 3A DLT assessment. Tolerability of zolbetuximab in combination with mFOLFOX6 and nivolumab in Japanese subject(s) will be evaluated in Cohort 4B, if Japanese subjects are not enrolled in the Cohort 4A DLT assessment.

ELIGIBILITY:
Inclusion Criteria:

* Female subject eligible to participate if she is not pregnant and at least one of the following conditions applies:

  * Not a woman of child-bearing potential (WOCBP) OR
  * WOCBP who agrees to follow the contraceptive guidance throughout the treatment period and for at least 9 months after the final oxaliplatin administration and 6 months after the final administration of all other study drugs.
* Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 6 months after the final study drug administration.
* Female subject must agree not to donate ova starting at screening and throughout the study period, and for 9 months after the final oxaliplatin administration and 6 months after the final administration of all other study drugs.
* A sexually active male subject with a female partner(s) who is of child-bearing potential must agree to use contraception during the treatment period and for at least 6 months after the final study drug administration.
* Male subject must agree not to donate sperm starting at screening and throughout the study period, and for 6 months after the final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study period and for 6 months after the final study drug administration.
* Subject has histologically confirmed gastric or GEJ adenocarcinoma.
* Cohorts 1-4: Subject has radiographically-confirmed, locally advanced, unresectable or metastatic disease within 28 days prior to the first dose of study treatment.
* Subject's tumor is positive for CLDN18.2 expression demonstrating moderate to strong membranous staining as determined by central IHC testing.
* Subject agrees to not participate in another interventional study while on treatment.
* Subject has ECOG performance status 0 to 1.
* Subject has predicted life expectancy ≥ 12 weeks.
* Subject must meet all of the following criteria based on the centrally or locally analyzed laboratory tests collected within 14 days prior to the first dose of study treatment. In case of multiple central laboratory data within this period, the most recent data should be used.

  * Hemoglobin (Hgb) ≥ 9 g/dL (transfusion is allowed, but post-transfusion Hgb [24 hours or later following transfusion] must be ≥ 9 g/dL)
  * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
  * Platelets ≥ 100 × 10^9/L
  * Albumin ≥ 2.5 g/dL
  * Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN in subjects without liver metastases (≤ 5 × ULN if liver metastases are present)
  * Cohorts 1-4: Estimated creatinine clearance ≥ 30 mL/min
  * Cohort 5: Serum creatinine ≤ 1.5 × ULN, or estimated creatinine clearance ≥ 50 mL/min for subjects with serum creatinine levels > 1.5 × ULN
  * Prothrombin time/international normalized ratio and partial thromboplastin time ≤ 1.5 × ULN (except for subjects receiving anticoagulation therapy)

Specific to Cohort 1A:

* Subject has measurable disease according to RECIST 1.1 within 28 days prior to the first dose of study treatment per investigator assessment. For subjects with only 1 evaluable lesion and prior radiotherapy ≤ 3 months before enrollment, the lesion must either be outside the field of prior radiotherapy or must have documented progression following radiation therapy.
* Subject has disease progression on or after at least 2 prior regimens for their advanced disease, including fluoropyrimidine and platinum-containing chemotherapy, and if appropriate, HER2/neu-targeted therapy and all associated side effects have resolved to grade 1 or less.
* Subject must have an additional available tumor specimen collected within 3 months prior to the first dose of study treatment.
* Subject must be an appropriate candidate for a tumor biopsy and is amenable to undergo a tumor biopsy during the screening period (if applicable) and treatment period as indicated in the Schedule of Assessments.

Specific to Cohort 2:

* Subject has measurable disease according to RECIST 1.1 within 28 days prior to the first dose of study treatment per investigator assessment. For subjects with only 1 evaluable lesion and prior radiotherapy ≤ 3 months before enrollment, the lesion must either be outside the field of prior radiotherapy or must have documented progression following radiation therapy.
* Subject has not received prior systemic anti-cancer therapy for their advanced disease (subject may have received neoadjuvant and/or fluorouracil-containing adjuvant chemotherapy as long as it has been completed ≥ 6 months before the first dose of study treatment).
* Subject has a gastric or GEJ tumor that is HER2-negative as determined by local or central testing.
* Subject must have an additional available tumor specimen collected within 3 months prior to the first dose of study treatment.
* Subject must be an appropriate candidate for a tumor biopsy and is amenable to undergo a tumor biopsy during the screening period (if applicable) and treatment period as indicated in the Schedule of Assessments.

Specific to Cohort 3A:

* Subject has radiologically evaluable disease (measurable and/or non-measurable) according to RECIST 1.1, per local assessment, ≤ 28 days prior to the first dose of study treatment. For subjects with only 1 evaluable lesion and prior radiotherapy ≤ 3 months before enrollment, the lesion must either be outside the field of prior radiotherapy or must have documented progression following radiation therapy.
* Subject has disease progression on or after at least 2 prior regimens for their advanced disease, including fluoropyrimidine and platinum-containing chemotherapy, and if appropriate, HER2/neu-targeted therapy.
* Subject has not received prior checkpoint inhibitor therapy.

Specific to Cohort 4A and 4B:

* Subject has radiologically evaluable disease.
* Subject has not received prior systemic anti-cancer therapy for their advanced disease.
* Subject has a gastric or GEJ tumor that is HER2-negative as determined by local or central testing.
* Subject has not received prior checkpoint inhibitor therapy.

Specific to Cohort 4B Only:

* Subject must have an additional available tumor specimen collected within 3 months prior to the first dose of study treatment.
* Subject must be an appropriate candidate for a tumor biopsy and is amenable to undergo a tumor biopsy during the screening period (if applicable) and treatment period.

Specific to Cohort 5 Only:

* Subject has new histologically confirmed primary gastric or GEJ adenocarcinoma that is amenable to curative resection.
* Subject has locoregional, resectable gastric or GEJ adenocarcinoma. GEJ may include type I-III Siewert classification. Clinical stage will be determined by endoscopic ultrasound (EUS) and/or CT or MRI. Diagnostic laparoscopy may be used as per institutional guidelines and clinical practices.
* Subject meets one of the following criteria of locoregional disease by clinical TNM staging:
* GEJ: cT2,N0 (high risk-lesions: ≥ 3 cm, poorly differentiated), cT1b-cT2,N+ or cT3-cT4a,Any N.
* Gastric: T2 to T4a, and/or N1-3,M0.
* Subject's tumor expresses CLDN18.2 in ≥ 75% of tumor cells demonstrating moderate to strong membranous staining as determined by central IHC testing

Exclusion Criteria:

* Subject has had prior severe allergic reaction or intolerance to known ingredients of zolbetuximab or other monoclonal antibodies, including humanized or chimeric antibodies.
* Subject has known immediate or delayed hypersensitivity or contraindication to any component of study treatment.
* Subject has received other investigational agents or devices concurrently or within 28 days prior to first dose of study treatment.
* Subject has received systemic immunosuppressive therapy, including systemic corticosteroids 14 days prior to first dose of study treatment.
* Subject has a complete gastric outlet syndrome or a partial gastric outlet syndrome with persistent recurrent vomiting.
* Subject has significant gastric bleeding and/or untreated gastric ulcers that would preclude the subject from participation.
* Subject has history of central nervous system metastases and/or carcinomatous meningitis from gastric/GEJ cancer.
* Subject has a known history of a positive test for human immunodeficiency virus (HIV) infection or known active hepatitis B (positive hepatitis B surface antigen [HBsAg]) or hepatitis C infection.
* Subject has had within 6 months prior to first dose of study treatment any of the following: unstable angina, myocardial infarction, ventricular arrhythmia requiring intervention or hospitalization for heart failure.
* Subject has active infection requiring systemic therapy that has not completely resolved within 7 days prior to the start of study treatment.
* Subject has active autoimmune disease that has required systemic treatment within the past 3 months prior to the start of study treatment.
* Subject has a clinically significant disease or co-morbidity that may adversely affect the safe delivery of treatment within this study or make the subject unsuitable for study participation.
* Subject has psychiatric illness or social situations that would preclude study compliance.
* Subject has had a major surgical procedure ≤ 28 days before start of study treatment.
* Subject is without complete recovery from a major surgical procedure ≤ 14 days before start of study treatment

  * Subject has received radiotherapy for locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma ≤ 14 days (Cohorts 1 and 3A) and ≤ 28 days (Cohorts 2 and 4A or 4B) prior to start of study treatment and has NOT recovered from any related toxicity.
  * Subject has another malignancy, for which treatment is required.
* Cohort 2, 4 and 5 Only, subject has any of the following:

  * Prior severe allergic reaction or intolerance to any component of mFOLFOX6 or FLOT chemotherapeutics in this study
  * Known dihydropyrimidine dehydrogenase deficiency (DPD).
  * Known peripheral neuropathy > Grade 1 (absence of deep tendon reflexes as the sole neurological abnormality does not render the subject ineligible).
  * Sinusoidal obstruction syndrome, formerly known as veno-occlusive disease, if present, should be stable or improving.
  * History of clinically significant ventricular arrhythmias.
  * QTc interval > 450 msec for male subjects; QTc interval > 470 msec for female subjects.
  * History or family history of congenital long QT syndrome.
  * Cardiac arrhythmias requiring anti-arrhythmic medications (Subjects with rate controlled atrial fibrillation for > 1 month prior to first dose of study treatment are eligible).
* Cohorts 3A, 4A and 4B Only, subject has any of the following:

  * Ongoing or previous autoimmune disease or interstitial lung disease, active diverticulitis or gastrointestinal ulcerative disease, or solid organ or stem cell transplant (for Cohort 4) or other uncontrolled or clinically significant medical disorders.
  * Type 1 diabetes mellitus, endocrinopathies stably maintained on appropriate replacement therapy or skin disorders (e.g., vitiligo, psoriasis, or alopecia) not requiring systemic treatment are allowed.
  * Known history of serious hypersensitivity reaction to a known ingredient of pembrolizumab or nivolumab.
* Cohort 4B Only: Subjects has microsatellite instability-high or mismatch repair deficient tumors.
* Cohort 5 Only, subject has either of the following:

  * Subject cannot undergo curative resection per the investigator's judgment
  * Subject meets the following criterion of locoregional disease by clinical TNM staging: cT1N0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) of zolbetuximab as a single agent by central review (Cohort 1) | Up to 3 months
  The ORR is defined as the proportion of participants with complete or partial objective response based on Response Evaluation Criteria in Solid Tumors (RECIST) V1.1 (assessed by an independent review committee (IRC)).

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of zolbetuximab: Area Under the Concentration-time Curve from the Time of Dosing Extrapolated to Time Infinity (AUCinf) (Cohorts 1A, 2, 3A, 4 and 5) | Up to 16 months
  AUCinf will be derived from the PK serum samples collected.
PK of zolbetuximab: Area Under the Concentration-time Curve from the Time of Dosing Extrapolated to Time Infinity Percentage (AUCinf (%extrap)) (Cohorts 1A, 2, 3A, 4 and 5) | Up to 16 months
  AUCinf (%extrap) will be derived from the PK serum samples collected.
PK of zolbetuximab: Area Under the Concentration-time Curve from the Time of Dosing Until the Last Measurable Concentration (AUClast) (Cohorts 1A, 2, 3A, 4 and 5) | Up to 16 months
  AUClast will be derived from the PK serum samples collected.
PK of zolbetuximab: Area Under the Concentration-Time Curve from the Time of Dosing to the Start of the Next Dosing Interval (AUCtau) (Cohorts 1A, 2, 3A, 4 and 5) | Up to 16 months
  AUCtau will be derived from the PK serum samples collected.
PK of zolbetuximab: Maximum Concentration (Cmax) (Cohorts 1A, 2, 3A, 4 and 5) | Up to 16 months
  Cmax will be derived from the PK serum samples collected.
PK of zolbetuximab: Concentration Immediately Prior to Dosing (Ctrough) (Cohorts 1A, 2, 3A, 4 and 5) | Up to 16 months
  Ctrough will be derived from the PK serum samples collected.
PK of zolbetuximab: Time of Maximum Concentration (Tmax) (Cohorts 1A, 2, 3A, 4 and 5) | Up to 16 months
  Tmax will be derived from the PK serum samples collected.
PK of zolbetuximab: Terminal Elimination Half-life (T1/2) (Cohorts 1A, 2, 3A, 4 and 5) | Up to 16 months
  T1/2 will be derived from the PK serum samples collected.
PK of zolbetuximab: Time of the last measurable concentration (Tlast) (Cohorts 1A, 2, 3A, 4 and 5) | Up to 16 months
  Tlast will be derived from the PK serum samples collected.
PK of zolbetuximab: Clearance (CL) (Cohorts 1A, 2, 3A, 4 and 5) | Up to 16 months
  CL will be derived from the PK serum samples collected.
PK of zolbetuximab: Volume of Distribution During the Terminal Phase (Vz) (Cohorts 1A, 2, 3A, 4 and 5) | Up to 16 months
  Vz will be derived from the PK serum samples collected.
PK of oxaliplatin: AUCinf (Cohort 2) | Up to 16 months
  AUCinf will be derived from the PK plasma samples collected.
PK of oxaliplatin: AUCinf (%extrap) (Cohort 2) | Up to 16 months
  AUCinf (%extrap) will be derived from the PK plasma samples collected.
PK of oxaliplatin: AUClast (Cohort 2) | Up to 16 months
  AUClast will be derived from the PK plasma samples collected.
PK of oxaliplatin: Cmax (Cohort 2) | Up to 16 months
  Cmax will be derived from the PK plasma samples collected.
PK of oxaliplatin: Tmax (Cohort 2) | Up to 16 months
  Tmax will be derived from the PK plasma samples collected.
PK of oxaliplatin: T1/2 (Cohort 2) | Up to 16 months
  T1/2 will be derived from the PK plasma samples collected.
PK of oxaliplatin: Tlast (Cohort 2) | Up to 16 months
  Tlast will be derived from the PK plasma samples collected.
PK of oxaliplatin: CL (Cohort 2) | Up to 16 months
  TL will be derived from the PK plasma samples collected.
PK of oxaliplatin: Vz (Cohort 2) | Up to 16 months
  Vz will be derived from the PK plasma samples collected.
PK of fluorouracil bolus (5-FU): AUCinf (Cohort 2) | Up to 16 months
  AUCinf will be derived from the PK plasma samples collected.
PK of fluorouracil bolus (5-FU): AUCinf (%extrap) (Cohort 2) | Up to 16 months
  AUCinf (%extrap) will be derived from the PK plasma samples collected.
PK of fluorouracil bolus (5-FU): AUClast (Cohort 2) | Up to 16 months
  AUClast will be derived from the PK plasma samples collected.
PK of fluorouracil bolus (5-FU): Cmax (Cohort 2) | Up to 16 months
  Cmax will be derived from the PK plasma samples collected.
PK of fluorouracil bolus (5-FU): Tmax (Cohort 2) | Up to 16 months
  Tmax will be derived from the PK plasma samples collected.
PK of fluorouracil bolus (5-FU): T1/2 (Cohort 2) | Up to 16 months
  T1/2 will be derived from the PK plasma samples collected.
PK of fluorouracil bolus (5-FU): Tlast (Cohort 2) | Up to 16 months
  Tlast will be derived from the PK plasma samples collected.
PK of fluorouracil bolus (5-FU): CL (Cohort 2) | Up to 16 months
  CL will be derived from the PK plasma samples collected.
PK of fluorouracil bolus (5-FU): Vz (Cohort 2) | Up to 16 months
  Vz will be derived from the PK plasma samples collected.
Safety and tolerability assessed by adverse events (AEs) (Cohorts 1A, 2, 3A, 4 and 5) | Up to 16 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Number of participants with electrocardiogram (ECG) abnormalities and or adverse events (Cohorts 1A, 2, 3A, 4 and 5) | Up to 14 months
  Number of participants with potentially clinically significant ECG values.
Number of participants with vital signs abnormalities and or adverse events (Cohorts 1A, 2, 3A, 4 and 5) | Up to 14 months
  Number of participants with potentially clinically significant vital sign values.
Number of participants with European Cooperative Oncology Group (ECOG) performance status abnormalities and or adverse events (Cohorts 1A, 2, 3A, 4 and 5) | Up to 14 months
  Number of participants with potentially clinically significant ECOG performance status values. ECOG grades 0-5, where 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4 = Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair and 5 = Dead.
Number of participants with laboratory assessments abnormalities and or adverse events (Cohorts 1A, 2, 3A, 4 and 5) | Up to 14 months
  Number of participants with potentially clinically significant laboratory values.
Number of anti-drug antibody (ADA) Positive Participants (Cohorts 1A, 2, 3A, 4 and 5) | Up to 16 months
  Immunogenicity will be measured by the number of participants that are ADA positive.
Health Related Quality of Life (HRQoL) measured by the Quality of Life Questionnaire - Core Questionnaire (QLQ-C30) questionnaire (Cohorts 1A, 2, 3A, 4 and 5) | Up to 16 months
  The EORTC-QLQ-C30 is a cancer-specific instrument consisting of 5 functional domain scales: physical, role, emotional, social and cognitive.
HRQoL measured by the Oesophago-Gastric Module (EORTC QLQ-OG-25) questionnaire (Cohorts 1A, 2, 3A, 4 and 5) | Up to 16 months
  The EORTC-QLQ-OG25 instrument evaluates GC- and GEJC-specific symptoms such as stomach discomfort, difficulties eating and swallowing and indigestion.
HRQoL measured by the Global Pain (GP) questionnaire (Cohorts 1A, 2, 3A, 4 and 5) | Up to 16 months
  The GP instrument is a single assessment of overall pain.
HRQoL measured by the EuroQOL Five Dimensions Questionnaire 5L (EQ-5D-5L) questionnaire (Cohorts 1A, 2, 3A, 4 and 5) | Up to 16 months
  The EQ-5D-5L is a standardized instrument developed by the EuroQol Group for use as a generic, preference-based measure of health outcomes. The EQ-5D-5L is a 5-item self-reported measure of functioning and wellbeing, which assesses 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension comprises 5 levels (no problems, slight problems, moderate problems, severe problems, extreme problems). A unique EQ-5D-5L health state is defined by combining 1 level from each of the 5 dimensions. This questionnaire also records the respondent's self-rated health status on a vertical graduated (0 = the worst health a participant can imagine to 100 = the best health a participant can imagine) visual analogue scale. Responses to the 5 items will also be converted to a weighted health state index (utility score) based on values derived from general population samples.
HRQoL measured by the Health Resource Utilization (HRU) questionnaire (Cohorts 1A, 2, 3A, 4 and 5) | Up to 16 months
  Health resource utilization questionnaire to assess the number of office visits, hospital stays and other healthcare resource utilization that occur outside of the clinical trial.
Disease Control Rate (DCR) of zolbetuximab as a single agent by investigator assessment (Cohort 1A) | Up to 3 months
  The DCR is defined as the proportion of subjects with complete or partial objective response, or stable disease based on RECIST V1.1.
DCR of zolbetuximab in combination with mFOLFOX6 by investigator assessment (Cohort 2) | Up to 13 months
  The DCR is defined as the proportion of subjects with complete or partial objective response, or stable disease based on RECIST V1.1.
DCR of zolbetuximab in combination with mFOLFOX6 (with nivolumab) by investigator assessment (Cohort 4) | up to 13 months
  DCR is defined as the proportion of subjects with complete or partial objective response, or stable disease based on RECIST V1.1.
DCR of zolbetuximab as a single agent by independent central reader (Cohort 1A) | Up to 3 months
  The DCR is defined as the proportion of subjects with complete or partial objective response, or stable disease based on RECIST V1.1.
DCR of zolbetuximab in combination with mFOLFOX6 by Independent central reader (Cohort 2) | Up to 13 months
  The DCR is defined as the proportion of subjects with complete or partial objective response, or stable disease based on RECIST V1.1.
Duration of Response (DOR) of zolbetuximab as a single agent by investigator assessment (Cohort 1A) | Up to 3 months
  DOR is defined as the time from the date of the first response CR/PR (whichever is first recorded) to the date of radiographical progression/death or date of censoring.
DOR of zolbetuximab in combination with mFOLFOX6 by investigator assessment (Cohort 2) | Up to 13 months
  DOR is defined as the time from the date of the first response CR/PR (whichever is first recorded) to the date of radiographical progression/death or date of censoring.
DOR of zolbetuximab in combination with mFOLFOX6 (with nivolumab) by investigator assessment (Cohort 4) | up to 13 months
  DOR is defined as the time from the date of the first response CR/PR (whichever is first recorded) to the date of radiographical progression/death or date of censoring.
DOR of zolbetuximab as a single agent by independent central reader (Cohort 1A) | Up to 3 months
  DOR is defined as the time from the date of the first response CR/PR (whichever is first recorded) to the date of radiographical progression/death or date of censoring.
DOR of zolbetuximab in combination with mFOLFOX6 by independent central reader (Cohort 2) | Up to 13 months
  DOR is defined as the time from the date of the first response CR/PR (whichever is first recorded) to the date of radiographical progression/death or date of censoring.
Progression Free Survival (PFS) of zolbetuximab as a single agent by investigator assessment (Cohort 1A) | Up to 3 months
  PFS is defined as the time from date of treatment start until the date of radiological disease progression assessed by independent radiographic reviewer (IRR), or until death due to any cause.
PFS of zolbetuximab in combination with mFOLFOX6 by investigator assessment (Cohort 2) | Up to 13 months
  PFS is defined as the time from date of treatment start until the date of radiological disease progression assessed by independent radiographic reviewer (IRR), or until death due to any cause.
PFS of zolbetuximab in combination with mFOLFOX6 (with nivolumab) by investigator assessment (Cohort 4) | up to 13 months
  PFS is defined as the time from date of treatment start until the date of radiological disease progression assessed by independent radiographic reviewer (IRR), or until death due to any cause.
PFS of zolbetuximab as a single agent by independent central review (Cohort 1A) | Up to 3 months
  PFS is defined as the time from date of treatment start until the date of radiological disease progression assessed by independent radiographic reviewer (IRR), or until death due to any cause.
PFS of zolbetuximab in combination with mFOLFOX6 by independent central review (Cohort 2) | Up to 13 months
  PFS is defined as the time from date of treatment start until the date of radiological disease progression assessed by independent radiographic reviewer (IRR), or until death due to any cause.
ORR of zolbetuximab as a single agent by investigator assessment (Cohort 1A) | Up to 3 months
  The ORR is defined as the proportion of subjects with complete or partial objective response based on RECIST V1.1.
ORR of zolbetuximab in combination with mFOLFOX6 by investigator assessment (Cohort 2) | Up to 13 months
  The ORR is defined as the proportion of subjects with complete or partial objective response based on RECIST V1.1.
ORR of zolbetuximab in combination with mFOLFOX6 (with nivolumab) by investigator assessment (Cohort 4) | up to 13 months
  The ORR is defined as the proportion of subjects with complete or partial objective response based on RECIST V1.1.
ORR of zolbetuximab in combination with mFOLFOX6 by independent central reader (Cohort 2) | Up to 13 months
  The ORR is defined as the proportion of subjects with complete or partial objective response based on RECIST V1.1.
ORR of zolbetuximab in combination with pembrolizumab by independent central reader (Cohort 3A) | Up to 5 months
  The ORR is defined as the proportion of subjects with complete or partial objective response based on RECIST V1.1.
Overall Survival (OS) of zolbetuximab as a single agent (Cohort 1A) | Up to 7 months
  OS is defined as the time from the date of treatment start until the documented date of death from any cause.
OS of zolbetuximab in combination with mFOLFOX6 and nivolumab (Cohort 4B) | up to 56 Months
  OS is defined as the time from the date of treatment start until the documented date of death from any cause.
OS of zolbetuximab in combination with FLOT (Cohort 5) | Up to 72 months
  OS is defined as the time from the date of treatment start until the documented date of death from any cause.
Percentage of participants with surgical complications (Cohort 5) | Up to 8 months
  Percentage of participants with surgical complications will be reported.
Percentage of participants with surgical mortality as defined by death within 30 days of surgery (Cohort 5) | Up to 30 days
  Percentage of participants with surgical mortality as defined by death within 30 days of surgery will be reported.
Percentage of participants able to complete preoperative chemotherapy (Cohort 5) | Up to 2 months
  Percentage of participants able to complete preoperative chemotherapy will be reported.
Percentage of participants with perioperative mortality and morbidity at 30 days and 90 days post last dose (Cohort 5) | Up to 3 months
  Percentage of participants with perioperative mortality and morbidity at 30 days and 90 days post last dose will be reported.
Percentage of participants able to start postoperative chemotherapy (Cohort 5) | Up to 7 months
  Percentage of participants able to start postoperative chemotherapy will be reported.
Percentage of participants able to complete postoperative chemotherapy (Cohort 5) | Up to 9 months
  Percentage of participants able to complete postoperative chemotherapy will be reported.
Percentage of participants with radiological response at restaging (Cohort 5) | Up to 5 months
  Radiological response will include complete response and partial response.
Percentage of subjects with pathological response (ypTNM) (Cohort 5) | Up to 5 months
  Pathological response (ypTNM) will include ypCR, ypPR
Disease-free Survival (DFS) (Cohort 5) | Up to 70 months
  DFS is defined as the time from date of treatment start until the date of radiological disease recurrence or until death due to any cause, whichever is earliest.
Minimal Residual Disease (Cohort 5) | Up to 37 months
  Minimal residual disease and disease recurrence as measured by circulating tumor DNA (ctDNA) will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Lead, Study Director — Astellas Pharma Global Development, Inc.
Locations (21):
- United States (6):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - UCLA Medical Center, Santa Monica, California
  - University of Chicago, Chicago, Illinois
  - Mass General / North Shore Can, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
- France (4):
  - Site FR33003, Pessac, Nouvelle-Aquitaine
  - Site FR33002, Poitiers, Nouvelle-Aquitaine
  - Site FR33001, Brest
  - Site FR33004, Paris
- Italy (4):
  - Site IT39005, Milan
  - Site IT39002, Napoli
  - Site IT39004, Padua
  - Site IT39003, Pisa
- Japan (3):
  - Site JP81001, Chiba
  - Site JP81002, Tokyo
  - Site JP81003, Tokyo
- South Korea (2):
  - Site KR82002, Seongnam-si
  - Site KR82001, Seoul
- Taiwan (2):
  - Site TW88601, Taichung
  - Site TW88602, Tainan

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/